CLINICAL TRIAL: NCT05965804
Title: Muscle Activation Patterns During the McMurray's Test for Knee Examination
Brief Title: Vastus Medialis Activation During McMurray's Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: PT-VMM-001
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Electromyography; Knee Injuries; Knee Pain Chronic
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adults: 30 healthy adult participants aged 18-45 years performing the McMurray knee examination test
  Interventions: Diagnostic Test: McMurray knee examination test

INTERVENTIONS:
Diagnostic Test: McMurray knee examination test — The McMurray test will be performed in different knee flexion and rotation angles.

SUMMARY:
This study will use electromyography to evaluate activation patterns of the vastus medialis and vastus lateralis muscles during the McMurray's knee examination test in different knee positions.

DETAILED DESCRIPTION:
The McMurray test is commonly used to assess knee pathology. However, it is unclear which knee position during this test best isolates activity of the vastus medialis muscle. This study will measure vastus medialis and lateralis activation using surface electromyography in 30 healthy participants performing the McMurray test. Different knee flexion and rotation angles will be evaluated to determine which position optimally activates the vastus medialis. Results may enhance utilization of the McMurray test in rehabilitation programs targeting this muscle.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-45 years
* No history of knee pathology

Exclusion Criteria:

* Contraindications to EMG
* Neurological or muscular disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy men and women aged 18-45 recruited from the local community.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-07-25 (Estimated); Primary Completion 2023-11-25 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Vastus Medialis Activation | Baseline
  Mean EMG activity of the vastus medialis during McMurray test at different knee positions. Measured in microvolts (μV).

SECONDARY OUTCOMES:
Vastus lateralis EMG activity during McMurray test (μV) | baseline
  Mean EMG activity of the vastus lateralis muscle during the McMurray knee examination test at different knee flexion and rotation angles. Measured in microvolts (μV).
Force exerted during McMurray test measured by dynamometer (Newtons) | baseline
  Maximum voluntary isometric knee extension force measured using a handheld dynamometer during the McMurray knee examination test at different knee positions. Measured in Newtons (N).

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No